CLINICAL TRIAL: NCT01756157
Title: A Phase 2, Randomized, Double-Blind, Multicenter, Dose-Ranging, Crossover Study to Evaluate the Safety and Efficacy of Subcutaneous Administration of CINRYZE® (C1 Esterase Inhibitor [Human]) With Recombinant Human Hyaluronidase (rHuPH20) for the Prevention of Angioedema Attacks in Adolescents and Adults With Hereditary Angioedema
Brief Title: Subcutaneous CINRYZE With Recombinant Human Hyaluronidase for Prevention of Angioedema Attacks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0624-206; 2012-000083-24 (EudraCT Number)
Record Dates: First submitted 2012-06-29; First posted 2012-12-25 (Estimated); Results first posted 2015-06-12 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: Crossover; C1 esterase inhibitor; Prevention; C1 inhibitor; Hereditary Angioedema; Subcutaneous; Recombinant human hyaluronidase
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — SERPING1 protein, human; Complement C1 Inhibitor Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SC CINRYZE with rHuPH20 Dose Level 1 followed by Dose Level 2 (Experimental): SC CINRYZE with rHuPH20 Dose Level 1 twice weekly (every 3 or 4 days) for 8 weeks followed by SC CINRYZE with rHuPH20 Dose Level 2 twice weekly (every 3 or 4 days) for 8 weeks.
  Interventions: Biological: CINRYZE with rHuPH20
- SC CINRYZE with rHuPH20 Dose Level 2 followed by Dose Level 1 (Experimental): SC CINRYZE with rHuPH20 Dose Level 2 twice weekly (every 3 or 4 days) for 8 weeks followed by SC CINRYZE with rHuPH20 Dose Level 1 twice weekly (every 3 or 4 days) for 8 weeks.
  Interventions: Biological: CINRYZE with rHuPH20

INTERVENTIONS:
Biological: CINRYZE with rHuPH20
  Other Names: C1 esterase inhibitor (human); Recombinant human hyaluronidase

SUMMARY:
The primary objectives of the study are to evaluate the safety, tolerability, and efficacy of two doses of CINRYZE with recombinant human hyaluronidase (rHuPH20) administered by subcutaneous (SC) injection to prevent angioedema attacks.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥12 years of age.
* Have a confirmed diagnosis of Hereditary Angioedema.

Exclusion Criteria:

* Receipt of any C1 inhibitor (C1 INH) therapy or any blood products for treatment or prevention of an angioedema attack within 7 days before the first dose of study drug.
* Be receiving prophylactic intravenous CINRYZE that exceeds 1000 units every 3 or 4 days (maximum weekly dose 2000 units).
* Have received any androgen therapy (e.g., danazol, oxandrolone, stanozolol, testosterone) within 7 days prior to the first dose of study drug.
* If female, have started taking or changed the dose of any hormonal contraceptive regimen or hormone replacement therapy (i.e., estrogen/progestin containing products) within 3 months prior to the first dose of study drug.
* History of allergic reaction to C1 INH products, including CINRYZE or other blood products.
* History of abnormal blood clotting.
* Have a known allergy to hyaluronidase or any other ingredient in the study formulation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-02-04 (Actual); Primary Completion 2013-09-13 (Actual); Study Completion 2013-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (23):
- United States (17):
  - ViroPharma Investigational Site, Birmingham, Alabama
  - ViroPharma Investigational Site, Scottsdale, Arizona
  - ViroPharma Investigational Site, Bentonville, Arkansas
  - ViroPharma Investigational Site, Walnut Creek, California
  - ViroPharma Investigational Site, Colorado Springs, Colorado
  - ViroPharma Investigational Site, Tampa, Florida
  - ViroPharma Investigational Site, Boston, Massachusetts
  - ViroPharma Investigational Site, Las Vegas, Nevada
  - ViroPharma Investigational Site, Mineola, New York
  - ViroPharma Investigational Site, Cincinnati, Ohio
  - ViroPharma Investigational Site, Columbus, Ohio
  - ViroPharma Investigational Site, Lake Oswego, Oregon
  - ViroPharma Investigational Site, Hershey, Pennsylvania
  - ViroPharma Investigational Site, Pittsburgh, Pennsylvania
  - ViroPharma Investigational Site, Knoxville, Tennessee
  - ViroPharma Investigational Site, Dallas, Texas
  - ViroPharma Investigational Site, Spokane, Washington
- Germany (4):
  - ViroPharma Investigational Site, Berlin
  - ViroPharma Investigational Site, Essen
  - ViroPharma Investigational Site, Mainz
  - ViroPharma Investigational Site, München
- ViroPharma Investigational Site, Barcelona, Spain
- ViroPharma Investigational Site, Jönköping, Sweden

REFERENCES:
- [Result] Riedl MA, Lumry WR, Li HH, Banerji A, Bernstein JA, Ba M, Bjrkander J, Magerl M, Maurer M, Rockich K, Chen H, Schranz J. Subcutaneous administration of human C1 inhibitor with recombinant human hyaluronidase in patients with hereditary angioedema. Allergy Asthma Proc. 2016 Nov;37(6):489-500. doi: 10.2500/aap.2016.37.4006. PMID 27931305
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 24 sites (United States=20, Europe=4) between 04 February 2013 (first participant dosed) and 13 September 2013 (last participant contact). Of 52 screened participants, 47 were randomized and treated. Screen failure reasons were consent withdrawn by 1 participant and violation of eligibility criteria by 4 participants.
Pre-assignment Details: Due to emergence of, and unexpected incidence and titer of, non-neutralizing anti-rHuPH20 antibodies in some subjects after administration of CINRYZE+rHuPH20, sponsor decided to stop dosing subjects with rHuPH20 and thus close the study. However, the study was completed with collection of safety data as outlined in the protocol.
Groups:
- Treatment Sequence A/B: Participants received Treatment A in Period 1 and Treatment B in Period 2; for 8 weeks each as a single 20 milliliter (mL) subcutaneous (SC) injection per dose. A washout period of at least 7 days and no more than 30 days was maintained between the last dose in Period 1 and the first dose in Period 2. Treatment A: 1000 U CINRYZE with 24,000 U rHuPH20 twice weekly (every 3 or 4 days) for 8 weeks. Treatment B: 2000 U CINRYZE with 48,000 U rHuPH20 twice weekly (every 3 or 4 days) for 8 weeks.
- Treatment Sequence B/A: Participants received Treatment B in Period 1 and Treatment A in Period 2; for 8 weeks each as a single 20 mL SC injection per dose. A washout period of at least 7 days and no more than 30 days was maintained between the last dose in Period 1 and the first dose in Period 2. Treatment B: 2000 U CINRYZE with 48,000 U rHuPH20 twice weekly (every 3 or 4 days) for 8 weeks. Treatment A: 1000 U CINRYZE with 24,000 U rHuPH20 twice weekly (every 3 or 4 days) for 8 weeks.
Period: First Intervention Period
Arm/Group | Treatment Sequence A/B | Treatment Sequence B/A
Started | 23 | 24
Completed | 22 | 22
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Period: Washout Period (at Least 7 Days)
Arm/Group | Treatment Sequence A/B | Treatment Sequence B/A
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0
Period: Second Intervention Period
Arm/Group | Treatment Sequence A/B | Treatment Sequence B/A
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat safety (ITT-S) population included all participants who received any amount of study drug.
Groups:
- Entire Study Population: Included participants who received 1000 U CINRYZE with 24,000 U rHuPH20 twice weekly (every 3 or 4 days) for 8 weeks (Treatment A) first and 2000 U CINRYZE with 48,000 U rHuPH20 twice weekly (every 3 or 4 days) for 8 weeks (Treatment B) first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Normalized Number of Angioedema Attacks During the Treatment Period
Description: Angioedema attack was defined as the participant-reported indication of symptoms or signs such as swelling or pain at any location following a report of no swelling or pain on the previous day. Manifestations of an attack that progress from one site to another, prior to complete resolution, was considered a single attack. Attacks that began to regress and then worsened before complete resolution was also considered one attack. Participants who were dosed but did not have any attacks in the period were assigned a value of zero. The number of attacks was normalized for the number of days participants participated in a given period and expressed as the monthly frequency.
Time Frame: From Visit 1 (Week 1) up to Visit 16 (Week 8) during each treatment period
Population: Intent-to-treat efficacy (ITT-E) population included all participants who completed both randomized treatment periods and fulfilled a priori defined evaluability criteria.
Measure: Mean (95% Confidence Interval); unit: angioedema attacks
Groups:
- Treatment A (1000 U CINRYZE + 24000 U rHuPH20): Participants received Treatment A (1000 U CINRYZE with 24,000 U rHuPH20 twice weekly [every 3 or 4 days] for 8 weeks) as a single 20 mL SC injection per dose in each treatment period.
- Treatment B (2000 U CINRYZE + 48000 U rHuPH20): Participants received Treatment B (2000 U CINRYZE with 48,000 U rHuPH20 twice weekly [every 3 or 4 days] for 8 weeks) as a single 20 mL SC injection per dose in each treatment period.
Arm/Group | Treatment A (1000 U CINRYZE + 24000 U rHuPH20) | Treatment B (2000 U CINRYZE + 48000 U rHuPH20)
Number analyzed (Participants) | 22 | 22
angioedema attacks | 1.58 [0.88 to 2.29] | 0.97 [0.41 to 1.53]
Statistical Analysis 1: Comparison: Treatment A (1000 U CINRYZE + 24000 U rHuPH20) vs Treatment B (2000 U CINRYZE + 48000 U rHuPH20); Test type: Superiority or Other; p = 0.0523, Paired t-test, 2 sided; Mean difference = -0.61, 95% CI 2-sided [-1.23 to 0.01]

2. Secondary Outcome: Cumulative Attack-severity During the Treatment Period
Description: Cumulative Attack-severity score was the sum of maximum symptom severity recorded for each angioedema attack, determined on the last day of symptoms and recorded as None=0, Mild=1, Moderate=2, and Severe=3 and summing over the unique attacks, yields a Cumulative Attack-severity score. None: no angioedema attack symptom; Mild: the angioedema attack symptom was noticeable to the participant but was easily tolerated and did not interfere with routine activities; Moderate: the angioedema attack symptom interfered with work/school or the ability to participate in family life and social activities; Severe: the angioedema attack symptom significantly limited the participant's ability to attend work/school or participate in family life and social activities. Cumulative attack-severity was normalized for the number of days participants participated in a given period and expressed as the monthly frequency. The scores ranged from 0 to 168 and higher scores represent worse symptoms.
Time Frame: From Visit 1 (Week 1) up to Visit 16 (Week 8) during each treatment period
Population: ITT-E population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Treatment A (1000 U CINRYZE + 24000 U rHuPH20) | Treatment B (2000 U CINRYZE + 48000 U rHuPH20)
Number analyzed (Participants) | 22 | 22
Score on a scale | 3.14 (3.79) | 1.81 (2.55)

3. Secondary Outcome: Cumulative Daily-severity During the Treatment Period
Description: Cumulative Daily-severity score was the sum of the severity scores recorded for every day of reported symptoms during the treatment period. Severity scores were recorded as None=0, Mild=1, Moderate=2, and Severe=3. None: no angioedema attack symptom; Mild: the angioedema attack symptom was noticeable to the participant but was easily tolerated and did not interfere with routine activities; Moderate: the angioedema attack symptom interfered with work/school or the ability to participate in family life and social activities; Severe: the angioedema attack symptom significantly limited the participant's ability to attend work/school or participate in family life and social activities. Cumulative daily severity was normalized for the number of days participants participated in a given period and expressed as the monthly frequency. The scores ranged from 0 to 168 and higher scores represent worse symptoms.
Time Frame: From Visit 1 (Week 1) up to Visit 16 (Week 8) during each treatment period
Population: ITT-E population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Treatment A (1000 U CINRYZE + 24000 U rHuPH20) | Treatment B (2000 U CINRYZE + 48000 U rHuPH20)
Number analyzed (Participants) | 22 | 22
Score on a scale | 4.63 (5.79) | 2.81 (4.42)

4. Secondary Outcome: Cumulative Symptomatic Days During the Treatment Period
Description: Cumulative symptomatic days was defined as the sum of the symptomatic days of each angioedema attack reported during the treatment period. Participants who were dosed but did not have any attacks in the period were assigned a value of zero. Cumulative symptomatic days was normalized for the number of days participants participated in a given period and expressed as the monthly frequency.
Time Frame: From Visit 1 (Week 1) up to Visit 16 (Week 8) during each treatment period
Population: ITT-E population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment A (1000 U CINRYZE + 24000 U rHuPH20) | Treatment B (2000 U CINRYZE + 48000 U rHuPH20)
Number analyzed (Participants) | 22 | 22
days | 3.06 (3.51) | 2.14 (3.30)

5. Secondary Outcome: Number of Angioedema Attacks Requiring Acute Treatment During the Treatment Period
Description: as for outcome 1
Time Frame: From Visit 1 (Week 1) up to Visit 16 (Week 8) during each treatment period
Population: ITT-E population
Measure: Mean (Standard Deviation); unit: angioedema attacks
Arm/Group | Treatment A (1000 U CINRYZE + 24000 U rHuPH20) | Treatment B (2000 U CINRYZE + 48000 U rHuPH20)
Number analyzed (Participants) | 22 | 22
angioedema attacks | 0.99 (1.51) | 0.43 (0.89)

ADVERSE EVENTS:
Time Frame: From the time of first dose of study drug up to 7 days after the last dose of study drug within each treatment period (8 weeks)
Description: Treatment-emergent adverse events included adverse events (AEs) that were not present at baseline (that is, prior to the first dose of study drug) but started during or after the first administration of study drug in each treatment period, and AEs that were present at baseline but worsened in frequency and/or severity. ITT-S population.
Arm/Group | Treatment A (1000 U CINRYZE + 24000 U rHuPH20) | Treatment B (2000 U CINRYZE + 48000 U rHuPH20)
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/46
Other Adverse Events (participants affected / at risk) | 42/44 | 46/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (1000 U CINRYZE + 24000 U rHuPH20) (N=44) | Treatment B (2000 U CINRYZE + 48000 U rHuPH20) (N=46)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hereditary angioedema (Congenital, familial and genetic disorders) | 32 (108) | 28 (69)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Injection site reactions (General disorders) | 37 (1113) | 40 (1212)
Injection site extravasation (General disorders) | 4 (15) | 9 (32)
Fatigue (General disorders) | 4 (5) | 1 (1)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Injury associated with device (General disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
Results of efficacy endpoints (time to first angioedema attack, effects of C1 inhibitor and C4 levels on clinical outcome during treatment period) were not reported due to early termination of the study but later completed for safety data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicentre publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicentre Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.